CLINICAL TRIAL: NCT01898572
Title: Carotid Intimae-media Thickness (CIMT) and Carotid Plaque (CP) Presence as Risk Markers of Cardiovascular Disease at the Time of Type 2 Diabetes Diagnosis
Brief Title: Carotid Atherosclerosis In Newly Diagnosed Type 2 Individuals
Acronym: DIABIMCAP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Consorci d'Atenció Primària de Salut de l'Eixample (Other)
Responsible Party: Principal Investigator, Emilio Ortega Martínez de Victoria, Senior Endocrinologist, MD, PhD, Hospital Clinic of Barcelona
Other Study IDs: PI11-DIABIMCAP; PI11/01723 (Other Grant/Funding Number: PI11/01723 Instituto de Salud Carlos III)
Record Dates: First submitted 2013-07-10; First posted 2013-07-12 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Type II Diabetes Mellitus Without Mention of Complication
Keywords: Newly Diagnosed Type II Diabetes Mellitus; Carotid Intimae-media Thickness; Carotid Plaque; Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Newly diagnosed T2DM: Newly diagnosed T2DM with no CVD. Standard care.
  Interventions: Other: Standard care
- Control individuals: Control individuals matched by age, gender, dyslipidemia, hypertension and smoking habit. Standard care.
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Standard care — Newly T2DM and control individuals will be controlled by their family care physician following standard (clinical guidelines) care.

SUMMARY:
It has been hypothesized, based on recent trials, that only early intervention can reduce cardiovascular morbidity and mortality in individuals with type 2 diabetes (T2DM). This finding may imply that atherosclerosis at diabetes diagnosed, is either negligible, or at early, or non-advanced, still modifiable disease stage. However, sparse information is available regarding atherosclerosis prevalence and its characteristics at diabetes presentation. Furthermore, although cardiovascular disease (CVD) prevention is the major goal of treatment in T2DM, risk assessment tools, mostly based on traditional CV risk factors, lack of adequate specificity to identify individuals at higher risk. Therefore, non-invasive tests, such as carotid ultrasound, have been recommended to better define CV risk in several groups of individuals, including those with intermediate risk or with T2DM.

This clinical study aims to improve the investigators knowledge on cardiovascular disease (CVD) in subjects with newly diagnosed T2DM (NEWDM). The investigators hypothesis is that carotid ultrasound (carotid intimae media thickness [CIMT] and carotid plaque [CP]) will show a worse subclinical/preclinical CVD stage in NEWDM compared with non-diabetic (CONTROL) individuals. Moreover, carotid ultrasound will also identify T2DM individuals at a higher risk in whom intervention should be more intensive.

Because individuals with T2DM have a higher prevalence of several CV risk factors, NEWDM will be matched with CONTROL individuals, not only for age and sex (the main determinants of atherosclerosis), but also for known, treated hypertension and dyslipidemia, and smoking habit.

The investigators will study NEWDM and CONTROL individuals without clinical CVD. This is a cross-sectional and longitudinal (18 months of follow-up) case-control study. The main study variables will be carotid ultrasound derived variables. The main aims of the study are: 1) to investigate CIMT and CP prevalence differences between NEWDM and CONTROL subjects; 2) to characterize the subset of NEWDM subjects with a higher CIMT (≥ mean+1SD o ≥ P75th) or CP presence; and 3) to early characterize individuals in whom subclinical CVD worsens (CIMT progression ≥ mean + 1SD o ≥ P75th) even after standard (according to clinical guidelines) diabetes treatment.

DETAILED DESCRIPTION:
Hypothesis:

In a Mediterranean population, the investigators hypothesized that the CIMT and the presence of carotid plaque (CP):

1. Are higher in patients with newly diagnosed T2DM than in a control population before and after adjusting for cardiovascular risk factors,
2. Can identify subjects with T2DM with increased cardiovascular risk at the beginning of the disease, and,
3. Can identify subjects in whom subclinical cardiovascular disease progresses despite treatment of T2DM according to clinical practice.

Aims:

Primary objectives:

1. To investigate differences in CIMT and the presence of CP in subjects with NEWDM and a control population. Cross-sectional study.
2. To identify and characterize the subset of NEWDM subjects presenting an increased CIMT (greater than the mean + 1SD or ≥ P75th) or carotid plaque presence. Cross-sectional study
3. To early characterize individuals in whom subclinical CVD worsens (CIMT progression ≥ mean + 1SD o ≥ P75th) even after multifactorial treatment of diabetes according to guidelines. Longitudinal study design with repeated measures.

Secondary objectives:

1. To study the main determinants of CIMT and the CP presence in NEWDM subjects and a control population. In addition to the cardiovascular risk factors will be studied:

   1. association with Mediterranean diet biomarkers (serum and urine) and diet adherence (semiquantitative food frequency questionnaire)
   2. genetic determinants of CVD
2. To investigate the main determinants of progression of CIMT in subjects treated according to clinical practice guidelines
3. To investigate the association of baseline CIMT, its progression, and the presence of CP with clinical scores used to estimate cardiovascular risk. These scores are: REGICOR (Registre Gironí del Cor: the Gerona Heart Register), a calibrated Framingham Score for a Mediterranean population, low risk SCORE (Systematic Coronary Risk Evaluation), and the UKPDS (United Kingdom Prospective Diabetes Study) score (specific for T2DM).
4. To identify carotid plaque biomarkers by a metabolomic approach

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women older than 40 years and less than 75 years.
* Newly Diagnosed T2DM (NEWDM). NEWDM is a subject without previous history of diabetes who has laboratory evidence consistent with diabetes (American Diabetes Association) within the last year.

Exclusion criteria:

* Previous cardiovascular events such as, but not limited to, myocardial infarction, acute coronary syndrome or chronic stroke, peripheral arterial disease, or revascularization surgery in any territory.
* Congestive heart failure (class III-IV).
* Cancer of any kind (except basal cell or for cervical carcinoma insitu) unless disease free is documented in the past five years.
* Anemia or known coagulopathy.
* Serum creatinine greater than 1.5 mg / dl or MDRD (Modification of Diet in Renal Disease) equation <50.
* Any organ transplant (except cornea)
* Known HIV-positive, active tuberculosis, malaria, chronic viral hepatitis B or C, cirrhosis of any aetiology.
* Pregnant or gestational idea in the next 2-3 years to inclusion.
* History of alcohol dependence (or abusive consumption) or other drugs in the past five years.
* Psychiatric illness that would entail adherence problems.
* Participation in a clinical trial protocol or investigational drugs.
* Debilitating chronic illness or short life expectancy to prevent adherence or therapeutic intensification is not the goal of managing your diabetes.
* ECG signs of ischemic heart disease.
* Diabetes type 1 or anti-GAD antibody positive.

Control population will be excluded based on the same criteria.

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care area: 3 Primary care centers in the city center of Barcelona (Spain)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-01; Primary Completion 2015-04 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Carotid Plaque presence(CP) | Baseline
  To investigate CP prevalence differences between NEWDM and CONTROL subjects
Carotid Intima Media Thickness (CIMT) | Baseline
  Compound CIMT (common carotid, bulb and internal carotid) differences between NEWDM and CONTROL.

SECONDARY OUTCOMES:
Changes in plaque height | Baseline to 18 months
Changes in CIMT at different territories | Baseline to 18 months
Changes in lifestyle | Baseline to 18 months
  Mediterranean Diet adherence and physical activity (validated questionnaires)
CIMT | Baseline
  CIMT differences in different territories (common carotid, bulb and internal carotid) between NEWDM and CONTROL.

OTHER OUTCOMES:
Changes in fat intake | Baseline to 18 months
  Blood cell membrane fatty acid composition was measured by gas chromatography
Diet intake | Baseline
  Food frequency questionnaire Serum and urine biomarkers Blood cell membrane fatty acid composition

CONTACTS AND LOCATIONS:
Overall Officials: Emilio Ortega, MD, PhD, Principal Investigator — Hospital Clinic Barcelona (Spain)
Locations (1):
- Hospital Clinic of Barcelona, Barcelona, Catalonia, Spain

REFERENCES:
- [Background] Ray KK, Seshasai SR, Wijesuriya S, Sivakumaran R, Nethercott S, Preiss D, Erqou S, Sattar N. Effect of intensive control of glucose on cardiovascular outcomes and death in patients with diabetes mellitus: a meta-analysis of randomised controlled trials. Lancet. 2009 May 23;373(9677):1765-72. doi: 10.1016/S0140-6736(09)60697-8. PMID 19465231
- [Background] Emerging Risk Factors Collaboration; Sarwar N, Gao P, Seshasai SR, Gobin R, Kaptoge S, Di Angelantonio E, Ingelsson E, Lawlor DA, Selvin E, Stampfer M, Stehouwer CD, Lewington S, Pennells L, Thompson A, Sattar N, White IR, Ray KK, Danesh J. Diabetes mellitus, fasting blood glucose concentration, and risk of vascular disease: a collaborative meta-analysis of 102 prospective studies. Lancet. 2010 Jun 26;375(9733):2215-22. doi: 10.1016/S0140-6736(10)60484-9. PMID 20609967
- [Background] Nambi V, Chambless L, Folsom AR, He M, Hu Y, Mosley T, Volcik K, Boerwinkle E, Ballantyne CM. Carotid intima-media thickness and presence or absence of plaque improves prediction of coronary heart disease risk: the ARIC (Atherosclerosis Risk In Communities) study. J Am Coll Cardiol. 2010 Apr 13;55(15):1600-7. doi: 10.1016/j.jacc.2009.11.075. PMID 20378078
- [Background] Stork S, van den Beld AW, von Schacky C, Angermann CE, Lamberts SW, Grobbee DE, Bots ML. Carotid artery plaque burden, stiffness, and mortality risk in elderly men: a prospective, population-based cohort study. Circulation. 2004 Jul 20;110(3):344-8. doi: 10.1161/01.CIR.0000134966.10793.C9. Epub 2004 Jul 6. PMID 15238459
- [Background] Wagenknecht LE, Zaccaro D, Espeland MA, Karter AJ, O'Leary DH, Haffner SM. Diabetes and progression of carotid atherosclerosis: the insulin resistance atherosclerosis study. Arterioscler Thromb Vasc Biol. 2003 Jun 1;23(6):1035-41. doi: 10.1161/01.ATV.0000072273.67342.6D. Epub 2003 Apr 17. PMID 12702517
- [Background] Pencina MJ, D'Agostino RB Sr, Larson MG, Massaro JM, Vasan RS. Predicting the 30-year risk of cardiovascular disease: the framingham heart study. Circulation. 2009 Jun 23;119(24):3078-84. doi: 10.1161/CIRCULATIONAHA.108.816694. Epub 2009 Jun 8. PMID 19506114
- [Background] Holman RR, Paul SK, Bethel MA, Matthews DR, Neil HA. 10-year follow-up of intensive glucose control in type 2 diabetes. N Engl J Med. 2008 Oct 9;359(15):1577-89. doi: 10.1056/NEJMoa0806470. Epub 2008 Sep 10. PMID 18784090
- [Background] ADVANCE Collaborative Group; Patel A, MacMahon S, Chalmers J, Neal B, Billot L, Woodward M, Marre M, Cooper M, Glasziou P, Grobbee D, Hamet P, Harrap S, Heller S, Liu L, Mancia G, Mogensen CE, Pan C, Poulter N, Rodgers A, Williams B, Bompoint S, de Galan BE, Joshi R, Travert F. Intensive blood glucose control and vascular outcomes in patients with type 2 diabetes. N Engl J Med. 2008 Jun 12;358(24):2560-72. doi: 10.1056/NEJMoa0802987. Epub 2008 Jun 6. PMID 18539916
- [Background] Action to Control Cardiovascular Risk in Diabetes Study Group; Gerstein HC, Miller ME, Byington RP, Goff DC Jr, Bigger JT, Buse JB, Cushman WC, Genuth S, Ismail-Beigi F, Grimm RH Jr, Probstfield JL, Simons-Morton DG, Friedewald WT. Effects of intensive glucose lowering in type 2 diabetes. N Engl J Med. 2008 Jun 12;358(24):2545-59. doi: 10.1056/NEJMoa0802743. Epub 2008 Jun 6. PMID 18539917
- [Background] Greenland P, Alpert JS, Beller GA, Benjamin EJ, Budoff MJ, Fayad ZA, Foster E, Hlatky MA, Hodgson JM, Kushner FG, Lauer MS, Shaw LJ, Smith SC Jr, Taylor AJ, Weintraub WS, Wenger NK, Jacobs AK, Smith SC Jr, Anderson JL, Albert N, Buller CE, Creager MA, Ettinger SM, Guyton RA, Halperin JL, Hochman JS, Kushner FG, Nishimura R, Ohman EM, Page RL, Stevenson WG, Tarkington LG, Yancy CW; American College of Cardiology Foundation; American Heart Association. 2010 ACCF/AHA guideline for assessment of cardiovascular risk in asymptomatic adults: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2010 Dec 14;56(25):e50-103. doi: 10.1016/j.jacc.2010.09.001. No abstract available. PMID 21144964
- [Derived] Bujosa F, Herreras Z, Catalan M, Pinyol M, Lamuela-Raventos RM, Martinez-Huelamo M, Gilabert R, Jimenez A, Ortega E, Chiva-Blanch G. Total carotene plasma concentrations are inversely associated with atherosclerotic plaque burden: A post-hoc analysis of the DIABIMCAP cohort. Clin Nutr. 2023 Jul;42(7):1168-1174. doi: 10.1016/j.clnu.2023.05.005. Epub 2023 May 13. PMID 37230851